CLINICAL TRIAL: NCT00443924
Title: A Multi-Center, Double-Masked, Randomized, Placebo-Controlled, Ascending Dose Study of INS115644 Ophthalmic Solution in Subjects With Bilateral Ocular Hypertension or Early Primary Open Angle Glaucoma
Brief Title: Study of INS115644 Ophthalmic Solution in Subjects With Ocular Hypertension or Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P08645; 032-101
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
Keywords: Bilateral ocular hypertension or early primary open angle glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- 1 (Placebo Comparator): Arm 1
  Interventions: Drug: Placebo
- 2 (Experimental): Arm 2
  Interventions: Drug: INS115644 Ophthalmic Solution
- 3 (Experimental): Arm 3
  Interventions: Drug: INS115644 Ophthalmic Solution
- 4 (Experimental): Arm 4
  Interventions: Drug: INS115644 Ophthalmic Solution
- 5 (Experimental): Arm 5
  Interventions: Drug: INS115644 Ophthalmic Solution

INTERVENTIONS:
Drug: INS115644 Ophthalmic Solution — One drop of Concentration #1 in one eye and one drop of placebo in contralateral eye every 12 hours for three days
  Arms: 2
Drug: Placebo — One drop of placebo in each eye every 12 hours for three days
  Arms: 1
Drug: INS115644 Ophthalmic Solution — One drop of Concentration #2 in one eye and one drop of placebo in the contralateral eye every twelve hours for three days
  Arms: 3
Drug: INS115644 Ophthalmic Solution — One drop of Concentration #3 in one eye and one drop of placebo in the contralateral eye every twelve hours for three days
  Arms: 4
Drug: INS115644 Ophthalmic Solution — One drop of Concentration #4 in one eye and one drop of placebo in the contralateral eye every twelve hours for three days
  Arms: 5

SUMMARY:
The purpose of this trial is to evaluate the safety and tolerability of INS115644 Ophthalmic Solution in subjects with bilateral ocular hypertension or early primary open angle glaucoma and to investigate the intraocular pressure lowering effects of INS115644 Ophthalmic Solution.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of bilateral ocular hypertension or early primary open angle glaucoma
* Have best corrected visual acuity in both eyes of at least +0.5 or better
* Have normal endothelial cell counts and morphology

Exclusion Criteria:

* Are diagnosed with closed angle glaucoma, exfoliation syndrome or exfoliation glaucoma, and pigment dispersion or secondary glaucoma
* Have a history of any type of intraocular surgery, except for cataract surgery
* Have had cataract surgery within three months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 28 days
Changes in intraocular pressure | 28 days